CLINICAL TRIAL: NCT03254082
Title: Glycemic Response of Cooked Grains Including Sorghum
Brief Title: Glycemic Response of Sorghum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: United Sorghum Checkoff Program (Unknown)
Responsible Party: Principal Investigator, Mark D. Haub, Professor, Kansas State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KSUHML10_Sorg
Record Dates: First submitted 2015-09-02; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Blood Glucose
Keywords: sorghum health
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- F-1000 (fontanelle flour) (Experimental): Fontenel sorghum flour
  Interventions: Other: Glycemic response of F-1000
- Sumac (Experimental): Sumac sorghum flour
  Interventions: Other: Glycemic response to sumac sorghum flour
- Wheat (Experimental): Wheat flour
  Interventions: Other: Glycemic response to wheat flour
- MMR (Experimental): MMR cultivar of sorghum flour -- from MMR Genetics, a company that produces sorghum seed.
  Interventions: Other: Glycemic response to MMR sorghum flour
- Sucrose (Active Comparator): Table sugar
  Interventions: Other: Glycemic response to sucrose

INTERVENTIONS:
Other: Glycemic response of F-1000 — The intervention was to determine if different flours elicit similar or different (change from baseline) 2 hour glucose responses (e.g., similar to glycemic index) after eating.
  Other Names: Fontanelle flour
  Arms: F-1000 (fontanelle flour)
Other: Glycemic response to sumac sorghum flour — The intervention was to determine the two hour change from baseline glucose responses (e.g., similar to glycemic index) after consuming sumac sorghum flour as a gruel.
  Arms: Sumac
Other: Glycemic response to MMR sorghum flour — The intervention was to determine the two hour change from baseline glucose responses (e.g., similar to glycemic index) after consuming MMR sorghum flour as a gruel.
  Arms: MMR
Other: Glycemic response to wheat flour — The intervention was to determine the two hour change from baseline glucose responses (e.g., similar to glycemic index) after consuming wheat flour as a gruel.
  Arms: Wheat
Other: Glycemic response to sucrose — The intervention was to determine the two hour change from baseline glucose responses (e.g., similar to glycemic index) after consuming sugar (dissolved in water)
  Other Names: sugar
  Arms: Sucrose

SUMMARY:
Given the interest in gluten-free foods and discovering dietary means to prevent metabolic disorders, this study was designed to determine the glycemic responses of four (4) grains and flours (corn, rice, wheat, and sorghum). The grain products (gruel) will be eaten by subjects and blood glucose will be collected prior to and after eating over the course of two hours. A dextrose solution, dosed to provide a like amount of available carbohydrate, will serve as the control treatment.

DETAILED DESCRIPTION:
Gruel was formed via a 1:9 ratio of grain (30 g) to water (270 ml) and cooked until thickened by placing water and grain mixture in a beaker and placed in a hot water bath (cooked over a stove/heating unit). The gruel was allowed to cool for 3-5 minutes before eating. The consistency of the gruel was similar to oatmeal. Subjects had a resting blood sample collected for assessment of fasting blood glucose, then ate the gruel (or control sucrose, 22g) that was assigned for that day -- they returned for the other gruel meals or sucrose control determined by Latin Square randomization. Finger stick blood samples where then collected at 30, 60, 90, and 120 minutes after eating the gruel (or sucrose) began.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy with no known diseases

Exclusion Criteria:

* Known metabolic, cancer, cardiovascular disease/condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Before eating (time 0) and 30, 60, 90, and 120 minutes after eating to measure the change in blood glucose due to the different food.
  This is an acute (over 2 hours) trial to measure blood glucose (glycemic response) to food.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haub, PhD, Principal Investigator — Kansas State University